CLINICAL TRIAL: NCT07372560
Title: Pharmacometric Modeling of a Hospital Preparation of Nicardipine Hydrochloride Oral Solution at 2 mg/mL in Hypertensive Patients in Pediatric Hematology-oncology
Brief Title: Pharmacometric Modeling of a Hospital Preparation
Acronym: PEDIATENS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0354/OB; N° IDRCB : 2025-A01969-40 (Other: ANSM)
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Hypertensive Patients
Keywords: Pharmacometric modeling; hématologie-oncologie pédiatrique

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of 6 x 1 mL tubes of plasma via functional catheter for nicardipine assay (collection before dose #1, then 30 minutes, 2 hours, 4 hours, 8 hours, and 24 hours after dose #1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of the pharmacokinetic parameters of an oral formulation of nicardipine hydrochloride — These pharmacokinetic parameters aim to optimize the use of this preparation in the management of pediatric hypertension. The pharmacokinetic parameters are: the area under the curve (AUC), the apparent volume of distribution (Vd/F), the apparent clearance (Cl/F), the maximum concentration (Cmax), the time to reach this concentration (Tmax), the elimination constant (ke), the elimination half-life (t1/2), the apparent intercompartmental clearance (Q/F), the apparent central volume (Vc/F), and the apparent peripheral volume (Vp/F).
  This kinetic profile will be obtained using Monolix® software modeling with the results of validated blood sampling methods. A small blood volume (1 mL) is required for these samples, which are taken from children who previously had a central venous catheter inserted.

SUMMARY:
Pediatric prescribers are very often faced with a lack of suitable therapies, particularly oral ones. This represents a major public health problem and necessitates adjustments to dosage or pharmaceutical form using medications marketed for adults, some of which contain excipients that may be harmful to children. This creates risks of dilution errors, administration errors, and the occurrence of adverse effects. Hospital pharmacy technicians are called upon daily to provide appropriate treatment for children. However, although this activity is authorized (Public Health Code, Good Preparation Practices), pharmacokinetic/pharmacodynamic studies on these preparations are only exceptionally carried out. Indeed, only stability studies are required to determine the expiration date of the preparation. Thus, prescribers are left without the necessary information to choose the dosage and administration schedule. Pediatric dosages are extrapolated from those for adults without any certainty of the treatment's effectiveness.

DETAILED DESCRIPTION:
The pediatric hematology-oncology department wanted to include an oral form of nicardipine in its therapeutic arsenal. Nicardipine is a widely used antihypertensive drug for secondary hypertension, particularly that caused by corticosteroid use. This oral form is preferred for its flexibility in dosing, which is based on weight and blood pressure readings. A first formulation was developed in 2017 and subsequently optimized in terms of excipients and raw material availability, leading to a second formulation in 2021. Nicardipine oral solution has been routinely prepared, dispensed, and administered for many years. The lack of bibliographic data concerning the use of nicardipine in a pediatric population prevents us from understanding the pharmacokinetic (PK) parameters, which are nevertheless essential for optimizing the benefit/risk balance of the drug and for individualizing doses. This study aims to optimize the use of this preparation in the management of hypertension in pediatrics and to promote the benefits of this formulation. This study is valuable because it is situated within the context of the routine therapeutic management of a patient in the pediatric hematology-oncology department suffering from hypertension. It therefore does not entail any modification of the child's care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 to 15 years, male or female.
* Patients followed in pediatric hematology-oncology.
* Patients with a central venous catheter as part of their initial care and available for blood sampling.
* Patients with a prescription for oral nicardipine (oral solution) whose formulation and/or dosage is/are not compatible with the commercial form of Loxen® 20 mg, requiring preparation.
* Patients requiring oral administration of nicardipine every 8 hours (initial prescription or renewal).
* Patients covered by a social security scheme.
* Parents/guardians informed of the study and not objecting to their child's participation
* For minors old enough to understand: patients who have not objected to the research.

Exclusion Criteria:

* Patient n'ayant pas un schéma d'administration toutes les 8 heures.
* Hypersensibilité à la substance active.
* Antécédent d'allergie à l'un des excipients (polysorbate 80, hypromellose, saccharine sodique, sorbate de potassium, acide citrique, citrate de sodium, saccharose).
* Refus de participation de l'enfant, des parents ou du représentant légal.
* Inclusion de l'enfant dans un autre essai clinique, si des prélèvements sanguins supplémentaires sont également prévus, dans un délai de 7 jours.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children in pediatric hematology-oncology requiring nicardipine administration as part of their standard care whether or not they are nicardipine-naïve (switching from the intravenous form used for hypertensive emergencies to the oral form, or patients already receiving hospital-prepared nicardipine oral solution at 2 mg/mL)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters in the target population of an oral formulation of nicardipine hydrochloride prepared by the pharmaceutical technology unit of the pharmacy at the Rouen University Hospital (Area Under the Curve (AUC)). | 24 hours
  This kinetic profile will be obtained through modeling using Monolix® software and the results of validated assays of the samples. A small blood volume (1 mL) is required for these samples, which are taken from children who previously had a central venous catheter inserted.
Pharmacokinetic parameters in the target population of an oral formulation of nicardipine hydrochloride prepared by the pharmaceutical technology unit of the pharmacy at the Rouen University Hospital (apparent distribution volume (Vd/F)). | 24 hours
  This kinetic profile will be obtained through modeling using Monolix® software and the results of validated assays of the samples. A small blood volume (1 mL) is required for these samples, which are taken from children who previously had a central venous catheter inserted.
Pharmacokinetic parameters in the target population of an oral formulation of nicardipine hydrochloride prepared by the pharmaceutical technology unit of the pharmacy at the Rouen University Hospital (apparent clearance (Cl/F)). | 24 hours
  This kinetic profile will be obtained through modeling using Monolix® software and the results of validated assays of the samples. A small blood volume (1 mL) is required for these samples, which are taken from children who previously had a central venous catheter inserted.
Pharmacokinetic parameters in the target population of an oral formulation of nicardipine hydrochloride prepared by the pharmaceutical technology unit of the pharmacy at the Rouen University Hospital (maximum concentration (Cmax)). | 24 hours
  This kinetic profile will be obtained through modeling using Monolix® software and the results of validated assays of the samples. A small blood volume (1 mL) is required for these samples, which are taken from children who previously had a central venous catheter inserted.
Pharmacokinetic parameters in the target population of an oral formulation of nicardipine hydrochloride prepared by the pharmaceutical technology unit of the pharmacy at the Rouen University Hospital (time to reach this concentration (Tmax)). | 24 hours
  This kinetic profile will be obtained through modeling using Monolix® software and the results of validated assays of the samples. A small blood volume (1 mL) is required for these samples, which are taken from children who previously had a central venous catheter inserted.
Pharmacokinetic parameters in the target population of an oral formulation of nicardipine hydrochloride prepared by the pharmaceutical technology unit of the pharmacy at the Rouen University Hospital (elimination constant (ke)). | 24 hours
  This kinetic profile will be obtained through modeling using Monolix® software and the results of validated assays of the samples. A small blood volume (1 mL) is required for these samples, which are taken from children who previously had a central venous catheter inserted.
Pharmacokinetic parameters in the target population of an oral formulation of nicardipine hydrochloride prepared by the pharmaceutical technology unit of the pharmacy at the Rouen University Hospital (elimination half-life (t1/2)). | 24 hours
  This kinetic profile will be obtained through modeling using Monolix® software and the results of validated assays of the samples. A small blood volume (1 mL) is required for these samples, which are taken from children who previously had a central venous catheter inserted.
Pharmacokinetic parameters in the target population of an oral formulation of nicardipine hydrochloride prepared by the pharmaceutical technology unit of the pharmacy at the Rouen University Hospital (clairance inter-compartimentale apparente (Q/F)). | 24 hours
  This kinetic profile will be obtained through modeling using Monolix® software and the results of validated assays of the samples. A small blood volume (1 mL) is required for these samples, which are taken from children who previously had a central venous catheter inserted.
Pharmacokinetic parameters in the target population of an oral formulation of nicardipine hydrochloride prepared by the pharmaceutical technology unit of the pharmacy at the Rouen University Hospital (apparent central volume (Vc/F)). | 24 hours
  This kinetic profile will be obtained through modeling using Monolix® software and the results of validated assays of the samples. A small blood volume (1 mL) is required for these samples, which are taken from children who previously had a central venous catheter inserted.
Pharmacokinetic parameters in the target population of an oral formulation of nicardipine hydrochloride prepared by the pharmaceutical technology unit of the pharmacy at the Rouen University Hospital (apparent peripheral volume (Vp/F)). | 24 hours
  This kinetic profile will be obtained through modeling using Monolix® software and the results of validated assays of the samples. A small blood volume (1 mL) is required for these samples, which are taken from children who previously had a central venous catheter inserted.

SECONDARY OUTCOMES:
Describe the distribution of the residual concentration at 24 hours | 24 hours
  Evaluate the determination of the residual concentration of nicardipine hydrochloride at 24 hours.
Demographic parameters of the studied population: sex | 24 hours
  Evaluate the demographic parameters of the studied population: sex
Demographic parameters of the studied population: age | 24 hours
  Evaluate the demographic parameters of the studied population: age
Demographic parameters of the studied population: weight . | 24 hours
  Evaluate the demographic parameters of the studied population: weight.
Demographic parameters of the studied population: height. | 24 hours
  Evaluate the demographic parameters of the studied population : height.
Dosages of the studied population: dose/kg/8 hours. | 24 hours
  Collection and measurement of prescribed nicardipine dosages: dose/kg/8 hours
A mathematical model capable of predicting, through simulation, exposure to and the antihypertensive effects of nicardipine in this population. | 24 hours
  Measurement of blood pressure (systolic and diastolic) and heart rate using a monitor to propose a mathematical model of pharmacodynamic parameters
Tolerance to treatment | 24 hours
  Collection of adverse events reported to the Regional Pharmacovigilance Centre (CRPV) in the context of routine practice
Acceptability of treatment | 24 hours
  The acceptability of the oral solution (in the form of a visual analog scale) will be assessed at each of the 3 doses

CONTACTS AND LOCATIONS:
Overall Officials: Marine MC CAVELIER, Doctor, Study Director — University Rouen Hospital; Thomas TD DUFLOT, Doctor, Study Chair — University Rouen Hospital
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.